CLINICAL TRIAL: NCT00560378
Title: A Long-term, Open Label, Noncomparative Study to Evaluate the Safety of 0.1% Tacrolimus (FK506) Ointment for Treatment of Atopic Dermatitis
Brief Title: Long-term Safety of Protopic in Atopic Eczema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-06-21
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic; Eczema, Atopic
Keywords: Tacrolimus; Administration, topical; Drug safety; Adults; Children
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus Ointment 0.1% (Experimental)
  Interventions: Drug: Tacrolimus ointment 0.1%

INTERVENTIONS:
Drug: Tacrolimus ointment 0.1% — Topical
  Other Names: Protopic

SUMMARY:
Patients who have participated in previous studies with Tacrolimus ointment for atopic eczema are entitled to enter this four-year follow study to investigate the safety of treatment with Tacrolimus ointment 0.1%

DETAILED DESCRIPTION:
A long-term, multi-centre, open label, non-comparative phase III study in patients with atopic dermatitis. All centres in Europe which have participated or are still participating in the FG-506-06-12, FG-506-06-18 or FG-506-06-19, FG-506-06-22 or FG-506-06-23 studies will be offered a participation in the protocol. Only patients enrolled by those centres for the above mentioned studies, who have received at least one dose of study medication can be enrolled. Tacrolimus ointment 0.1% will be administered until clearance of the skin occurs. Treatment is restarted after signs and symptoms reoccur. Safety will be assessed from adverse events reported by the patient/parent/guardian or observed by the investigator at the site of application and elsewhere. The safety evaluation will include monitoring of routine hematology and serum chemistry parameters at Baseline/Day 1, Week 1, Month 6, Month 12, Month 18, Month 24, Month 30, Month 36, Month 42 and/or at the end of the study (End-of-Study Visit).

ELIGIBILITY:
Inclusion Criteria:

* Every patient who has participated in the FG-506-06-12, FG-506-06-18, FG-506-06-19, FG-506-06-22 or FG-506-06-23 study, and has received at least one dose of study medication
* Patient is likely to benefit from further treatment with Tacrolimus (FK506) ointment in the opinion of the investigator
* Patient has atopic dermatitis with Body surface involvement between 5% and 60% for patients with the age of 2 years to 15 years (not having reached their 16th birthday) and between 5% and 100% for patients with 16 years of age or older

Exclusion Criteria:

* Patient has an infection requiring treatment
* Patient is known to be HIV positive
* Patient has a systemic disease, including cancer or history of cancer or AIDS, which would contraindicate the use of Tacrolimus (FK506) ointment

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 1998-06; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 4 Years

SECONDARY OUTCOMES:
Haematology and biochemistry parameters and vital signs | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma GmbH
Locations (41):
- Brussels, Belgium
- Aarhus, Denmark
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- France (10):
  - Bordeaux
  - Brest
  - Gaël
  - Lyon
  - Nantes
  - Paris
  - Pessac
  - Quimper
  - Saint-Etienne
  - Tours
- Germany (9):
  - Bonn
  - Düsseldorf
  - Erlangen
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - München
  - Münster
  - Tübingen
- Szeged, Hungary
- Ireland (2):
  - Cork
  - Dublin
- Riga, Latvia
- Amsterdam, Netherlands
- Warsaw, Poland
- Spain (3):
  - Barcelona
  - Madrid
  - Seville
- United Kingdom (8):
  - Cardiff
  - Coventry
  - Lancaster
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Southhampton

REFERENCES:
- [Background] Reitamo S, Rustin M, Harper J, Kalimo K, Rubins A, Cambazard F, Brenninkmeijer EE, Smith C, Berth-Jones J, Ruzicka T, Sharpe G, Taieb A; 0.1% Tacrolimus Ointment Long-term Follow-up Study Group. A 4-year follow-up study of atopic dermatitis therapy with 0.1% tacrolimus ointment in children and adult patients. Br J Dermatol. 2008 Sep;159(4):942-51. doi: 10.1111/j.1365-2133.2008.08747.x. Epub 2008 Jul 15. PMID 18637898